CLINICAL TRIAL: NCT07246330
Title: Stratified Treatment in Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma Without Progression After Chemoimmunotherapy Induction Plus Concurrent Chemoradiotherapy: Toripalimab Consolidation vs observation--a Prospective, Randomized, Controlled Phase III Multicenter Study
Brief Title: Stratified Treatment in Unresectable Locally Advanced ESCC Without Progression After Chemoimmunotherapy Induction Plus CCRT: Toripalimab Consolidation vs observation--a Prospective, Randomized, Controlled Phase III Multicenter Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SELECTor
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 (Experimental)
  Interventions: Drug: Toripalimab
- A2 (No Intervention)
- B1 (Experimental)
  Interventions: Drug: Toripalimab
- B2 (No Intervention)

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240 mg, administered on the first day of each cycle, and a cycle of administration every 3 weeks
  Arms: A1; B1

SUMMARY:
This study is a prospective, randomized controlled, phase III multicenter trial. Its objectives are to explore the stratified application of consolidation immunotherapy after chemoimmunotherapy induction plus concurrent chemoradiotherapy, identify the potential beneficiary population of consolidation immunotherapy, and evaluate the efficacy and safety of consolidation immunotherapy.

The main participants are patients with unresectable locally advanced esophageal squamous cell carcinoma who have undergone 2-4 cycles of chemoimmunotherapy induction followed by concurrent chemoradiotherapy. Imaging assessment should be completed within 1-84 days after the end of chemoradiotherapy. Eligible patients meeting the inclusion and exclusion criteria will be divided into the CR/PR cohort and SD cohort based on treatment response, and receive the following treatments respectively:

CR/PR cohort: Patients with a response assessment of CR (Complete Response) or PR (Partial Response) will be randomly assigned at a 1:1 ratio to:

Toripalimab monotherapy maintenance group (Group A1) vs. Observation group (Group A2) (116 patients vs. 116 patients)

SD cohort: Patients with a response assessment of SD (Stable Disease) will be randomly assigned at a 1:1 ratio to:

Toripalimab monotherapy maintenance group (Group B1) vs. Observation group (Group B2) (54 patients vs. 54 patients) The medication dosage is as follows: Toripalimab 240mg, intravenous infusion on Day 1, every 3 weeks (Q3W). A total of 3 treatment cycles will be administered. Subsequent treatment continuation will be determined by the patient. If continued, treatment will proceed until the occurrence of disease progression (radiological progression confirmed by RECIST v1.1), intolerable toxicity, initiation of new antitumor therapy, voluntary withdrawal of the subject from the study, or the investigator's judgment that the subject needs to withdraw. The maximum duration of medication is 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, signed informed consent, good compliance with follow-up;
2. Aged 18-75 years (inclusive), male or female;
3. Clinically staged II-IVa unresectable (AJCC 8th ed.: cT1N2-3M0/cT2-4bN0-3M0) or IVb (supraclavicular lymph node metastasis only); the patient had no disease progression after 2-4 cycles of chemo-immunotherapy induction combined with concurrent chemoradiotherapy (CCRT). Patients receiving CCRT must meet the following criteria: Patients with inoperable tumors must have received at least 2 cycles of weekly regimen or 1 cycle of 3-week platinum-based chemotherapy combined with radical radiotherapy (50-64 Gy) and have no evidence of radiographic disease progression (according to RECISTv1.1) as compared to before and after radical concurrent chemoradiation;
4. ECOG PS 0-1;
5. Expected survival ≥3 months;
6. Fresh or archived tumor tissue samples within 6 months should be provided for biomarker analysis. The sample type is FFPE tumor tissue block or at least 10 unstained FFPE tumor tissue sections with a thickness of 3-5 μm. For patients who cannot provide tissue samples meeting the above requirements, the investigator should discuss and determine whether to enroll;
7. Adequate organ and bone marrow function defined as:

   1. ANC ≥1.5×10⁹/L;
   2. Platelets ≥100×10⁹/L;
   3. Hemoglobin ≥9g/dL;
   4. Serum albumin ≥2.8g/dL;
   5. Total bilirubin ≤1.5×ULN; ALT/AST/AKP ≤2.5×ULN;
   6. Serum creatinine ≤1.5×ULN or creatinine clearance ≥60mL/min (Cockcroft-Gault);
   7. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN [Patients receiving stable-dose anticoagulant therapy (e.g., low-molecular-weight heparin or warfarin) with an INR within the expected therapeutic range of the anticoagulant are eligible];
8. Females of childbearing potential: negative pregnancy test within 72h pre-first dose; contraception during study + 6 months post-last dose. Males with fertile partners: contraception during study + 6 months post-last dose.

Exclusion Criteria:

1. Any unresolved NCI CTCAE ≥ grade 2 toxicity following prior chemoradiotherapy. Patients with irreversible and controllable hearing loss are eligible;
2. Small cell carcinoma, adenocarcinoma, or mixed carcinoma components in histology;
3. Grade ≥ 2 peripheral neuropathy based on NCI CTCAEv5.0 criteria
4. Found to have a higher risk of esophageal fistula by clinical assessment or imaging studies, such as a past history or related symptoms of esophageal fistula, or infiltration of the primary tumor into the great vessels or trachea;
5. Patients with any history of active autoimmune diseases or autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); patients without any intervention after adults except vitiligo or recovered childhood asthma/allergy; patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes treated with stable doses of insulin can be included;
6. History of immunodeficiency, including positive HIV test, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation;
7. Patients with uncontrolled cardiac clinical symptoms or diseases, such as (1) NYHA II and above heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
8. Serious infection (CTCAE > grade 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging showed active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug need oral or intravenous antibiotics, but excluding the prophylactic use of antibiotics; through the history or CT examination found active pulmonary tuberculosis infection, or within 1 year before enrollment found active pulmonary tuberculosis infection history, or more than 1 year ago had active pulmonary tuberculosis infection history but no regular treatment of patients;
9. Known allergies, hypersensitivity, or contraindications to terdiplimumab or any of the components used in its formulation;
10. Diagnosis of any other malignancy before the first use of study drugs, except for those with a low risk of metastasis and death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ;
11. Pregnant or lactating women; fertile subjects are unwilling or unable to take effective contraceptive measures;
12. According to the investigator 's judgment, the patient has other factors that may cause the patient to be forced to terminate the study halfway, such as suffering from other serious diseases (including mental illness) requiring concomitant treatment, and recently combined with other serious diseases (such as myocardial infarction, cerebrovascular accident) considering the high risk of recurrence, severely abnormal laboratory test values, family or social factors, which may affect the patient' s safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
1 year Progress Free Survival (PFS) rate | 12 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 36 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Overall survival (OS) | 36 months
  OS is the length of time from the date of randomization until death from any cause
Objective response rate (ORR) | 24 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.